CLINICAL TRIAL: NCT07180017
Title: Use of Tools for Early Detection of Cerebral Palsy: A Survey of Turkish Pediatric Physical Therapists
Brief Title: A Survey of Turkish Pediatric Physical Therapists
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, Associate Professor, Kahramanmaras Sutcu Imam University
Other Study IDs: Survey of Turkish Pediatric PT
Record Dates: First submitted 2025-09-05; First posted 2025-09-18 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Palsy (CP); Survey; Detection; Pediatric Physiotherapy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: All pediatric physiotherapists working in different cities in Turkey, reached through social media under the leadership of the therapists of the Developmental Physiotherapy and Pediatric Rehabilitation Unit of Gazi University Department of Physiotherapy and Rehabilitation

SUMMARY:
CP encompasses a group of persistent disorders of movement and posture development resulting from injury to the developing brain. Thanks to preventive measures and advances in obstetric and neonatal care, the incidence and severity of CP are currently decreasing in some countries, and the use of early diagnosis guidelines or protocols in follow-up units highlights the potential for faster recovery. A 2017 clinical review of early diagnosis tools, published by a group of international experts with best practice recommendations, called for earlier diagnosis through timely use of recommended tools. The diagnosis of CP is typically made by a physician between 12 and 24 months of age, but in some cases, it is delayed until 42 months. Early identification of a high risk of CP relies on a combination of a detailed patient history, developmental assessment, a structured and validated neurological examination or neuromotor assessment, and brain imaging studies. Conversely, the accurate and early use of key tools for early diagnosis can allow for much earlier detection of CP in infants younger than or older than 5 months.According to international guidelines, infants at high risk of CP should be monitored. This monitoring should be conducted by an interdisciplinary team, including a neonatologist, pediatrician, pediatric neurologist, pediatric physiotherapist, speech-language-swallowing therapist, and special education specialist. Pediatric physiotherapists are a crucial part of this team for developmental follow-up and rehabilitation. Therefore, it is important that pediatric physiotherapists in our country have sufficient awareness in this field, are equipped with various training programs, and reach international standards. This allows them to provide early guidance to families at risk of CP, facilitate early diagnosis of CP, and initiate treatment.The aim of this study was to evaluate the use of early diagnostic assessment tools in pediatric physiotherapy practice in Turkey for infants aged 0-2 years at risk for cerebral palsy (CP). Best practice guidelines worldwide recommend the timely use of key assessment tools to reduce the age at which CP is diagnosed. In this context, a digital survey administered to pediatric physiotherapists in Spain, translated into Turkish with the necessary permissions, will be used to determine the awareness levels of physiotherapists in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* All literate pediatric physiotherapists between the ages of 25-50 working in different provinces in Turkey

Exclusion Criteria:

* Physiotherapists with no experience in pediatric physiotherapy

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All pediatric physiotherapists working in different cities in Turkey, reached through social media under the leadership of the therapists of the Developmental Physiotherapy and Pediatric Rehabilitation Unit of Gazi University Department of Physiotherapy and Rehabilitation
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Digital survey for pediatric physiotherapists(PTs) | DAY1
  A purpose-built digital survey consisting of 45 multiple-choice questions with five thematic sections. The survey used in this context will be a survey administered digitally to pediatric physiotherapists in Spain, translated into Turkish with the necessary permissions. This survey will be administered via Google Forms.

SECONDARY OUTCOMES:
Demographic Information | DAY1
  Sosyodemographic information of PTs will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: hatice adıgüzel tat, Associate Professor, Principal Investigator — Kahramanmaras Sutcu Imam University; umut apaydın, Asisstant Prof, Study Chair — Karadeniz Technic University; Sabiha Bezgin, Asisstant Prof, Study Chair — Mustafa Kemal University; Bulent Elbasan, Proffessor, Study Director — Gazi University
Locations (1):
- Kahramanmaraş Sütçü imam University, Kahramanmaraş, Onikişubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No